CLINICAL TRIAL: NCT03239275
Title: Evaluation of Labial Versus Lingual Biocreative Therapy for en Masse Retraction of Maxillary Anterior Teeth: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Bio-creative Therapy for En Masse Retraction of the Maxillary Anterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mais Medhat Sadek, Assistant lecturer, Department of Orthodontics, Faculty of Dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORD14-1D
Record Dates: First submitted 2017-07-31; First posted 2017-08-04 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: en masse retraction; biocreative therapy; class II; skeletal anchorage
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labial biocreative therapy group (Experimental): Upper six anterior teeth will be bonded (0.018-inch slot brackets), leveled and aligned until reaching 0.017*0.025 stainless steel archwire.
  Right and left bracket head mini-screw (1.6*8 mm) will be inserted under local anaesthetic into the inter-radicular space between upper second premolar and first molar at the level of mucogingival junction. Crimpable hooks (10 mm) will be crimped onto the archwire between the upper lateral incisor and canine. 200 grams retraction force will be applied using NiTi coil springs from the hooks to the minscrew on both sides. Overlay reverse curve 0.016*0.022 NiTi will be inserted posteriorly into the mini-screw and ligated anteriorly to the archwire in the midline.
  Interventions: Procedure: Biocreative therapy
- Lingual biocreative therapy group (Active Comparator): En masse retraction of the six anterior teeth was accomplished using a lingual retractor bonded on to the lingual surface of the 6 anterior teeth, C-palatal plate fixed near the median palatal suture with 3 micro-screws, and Nickel Titanium (Ni-Ti) closing coil springs to apply a force of 200 g per side (total 400 g) directly from the C-plate to the lingual retractor.
  Interventions: Procedure: Biocreative therapy

INTERVENTIONS:
Procedure: Biocreative therapy

SUMMARY:
The purpose of this study is to compare the effectiveness and efficiency of labial versus lingual biocreative therapy in achieving en masse retraction of the maxillary anterior teeth in subjects with class II malocclusion requiring upper first premolar extraction.

DETAILED DESCRIPTION:
1. Background:

   Maximum anchorage is commonly required in patients with severe protrusion. Conventional retraction by sliding mechanics in extraction cases have been associated with variable degrees of anchorage loss. Use of miniscrew for reinforcement of orthodontic anchorage has become increasingly popular in recent years. Miniscrews are convenient, save time, and do not require patient cooperation. However, sliding mechanics with direct anchorage from mini-screw can have several biomechanical drawbacks. The force used during retraction is not reciprocal, posteriorly it is negated by the miniscrew, not by teeth. As a result, either the entire arch or the anterior segment rotates around the center of resistance. These mechanics produce posterior open bite and anterior deep overbite. To avoid this problem, Chung et al, introduced the technique that minimizes side effects by replacing the posterior appliance segments with the partially osteointegrated C-implant. This system was called "biocreative therapy".

   With the bio-creative approach, true intrusion vectors on the anterior teeth can be applied without unwanted reactive forces affecting the posterior teeth, the posterior teeth are left intact.

   In Labial biocreative therapy type I, a 0.016 × 0.022-in stainless steel utility archwire is placed from the anterior segment into the implant tube, and gable bends are used to generate an anterior torque moment on the anterior segment of the teeth to provide bodily movement during en-masse retraction. On the other hand, in biocreative therapy type II, en masse anterior retraction is accomplished by applying retraction force via NiTi coil springs between an anterior retraction hook placed between the lateral incisor and the canine and the skeletal anchorage. An overlay intrusion arch wire is used to generate torque on the anterior segment of teeth; thereby various patterns of tooth movement can be obtained through the combination of intrusion force, retraction force, and length of the retraction hook. Location and management of the center of resistance (Cres) with respect to retraction force vectors is critical. The clinician should select the length of a power arm according to the desired type of tooth movement; controlled lingual crown tipping, root tipping, or bodily movement.

   Adult orthodontics is an increasing part of the orthodontic practice. However, adult patients are often annoyed by the appearance of labial brackets and tend to delay or avoid starting orthodontic treatment. Lingual orthodontics is a viable option for these patients as being "invisible orthodontic treatment". The disadvantages of lingual orthodontics include the excessive chair time, complicated bio-mechanics, patient discomfort, expensive lab procedures, and high material prices. However, several innovations have improved the use of lingual orthodontics, such as customized lingual brackets and two-dimensional lingual brackets that can be bonded directly. Nonetheless, the efficient control of anterior torque and intrusion during retraction continues to be a limiting challenge.

   Mini-implants placed on each side of the palate have been used in conjunction with lingual orthodontics to avoid uncontrolled tipping and the deepening of the anterior bite during en masse retraction. A lever arm is soldered to the main lingual arch wire. This moves the force vector apically and closer to the center of resistance, thereby allowing better control of torque during retraction. However, play within the slot allows some of the torque to be lost during retraction. In addition, unwanted canting of the occlusal plane may occur if bilateral mini-implants are not in the same horizontal plane, due to different force vectors generated during retraction. Moreover, the sliding mechanics may be adversely affected by friction within bracket slots and tubes, causing unwanted distalization of posterior teeth.

   Lingual Biocreative therapy for anterior retraction offers several advantages. En masse retraction of the maxillary anterior dentition is achieved using C-lingual retractor and C-palatal plate. The C-lingual retractor is bonded to the lingual surfaces of the upper six anteriors, providing excellent esthetics. The C-palatal plate is fixed near the median palatal suture with mini-implants. The upper posterior orthodontic appliances are not needed as anchorage for 3-dimensional retraction of the upper anteriors.

   Lingual biocreative therapy technique can be used to provide patients with esthetic treatment, excellent anchorage control offered by skeletal anchorage, rapid and controlled retraction, simplified orthodontic bio-mechanics, and avoiding unnecessary use of complex orthodontic devices. Posterior teeth are not disturbed by friction in the appliance.

   As the majority of research work related to biocreative therapy technique was mainly case reports, three-dimensional finite element analyses, and three retrospective studies using two-dimensional cephalometric data, and the fact that no studies; up to the time of this writing; compared the labial and lingual biocreative techniques, the idea of this study has aroused as to use the advanced technology of three-dimensional imaging to clinically evaluate and compare the effects of labial and lingual biocreative therapy for en masse retraction of the maxillary anterior teeth.
2. Research Hypothesis:

   The null hypothesis (H0) of this research is that there will be no statistically significant differences between labial and lingual biocreative therapy in the mean change in the upper incisor inclination after en masse retraction of the anterior teeth in subjects with class II malocclusion requiring upper first premolar extraction.
3. Objectives:

   The primary objective of this study is to determine if there will be statistically significant differences between labial and lingual biocreative therapy in the mean change in the upper incisor inclination after en masse retraction of the anterior teeth.

   Secondary objectives include:

   To compare between labial and lingual biocreative therapy regarding:
   * Changes in the soft tissue parameters including the nasolabial angle, inter-labial gap, and position of the upper and lower lips in the antero-posterior dimension; that would contribute to soft tissue profile correction.
   * Molar anchorage loss.
   * Patient satisfaction from treatment with either the labial or lingual biocreative therapy.
   * Vertical movement of the crown of the six maxillary anterior teeth.
   * Changes in the transverse dimension of the upper arch.
   * Skeletal measurements including the mean change in the position of point A from the Nasion perpendicular plane and change in the SNA angle.
   * Time duration required to complete the retraction phase.
4. Study design According to the norms of the CONSORT STATEMENT, this study will be clinical with intervention, in which the allocation of the subjects will be randomized (block randomization). This study will be parallel with blinding for the outcome assessors. The primary purpose of this study will be treatment.
5. Participants - Settings and locations where the data are collected The treatment will be performed in the outpatient clinics of Department of Orthodontics of Ain Shams University. This public university predominantly serves low-income population living in Cairo, Egypt. Data will be collected from January 2016 through November 2017.
6. Interventions Two groups will receive treatment. Group 1 will be treated with the labial biocreative therapy group until the achievement of normal overjet (1 to 3 mm).

Group 2 will be treated with lingual biocreative therapy group until the achievement of normal overjet (1 to 3 mm).

7a. Sample size Sample size calculation was based on the studies by Kim et al and Kim et al. For the labial group, a mean change in the upper incisor inclination to SN plane of 15.33 degrees, with a standard deviation of 6.85 was reported by Kim et al who compared pre-treatment cephalometric radiographs with those taken after en-masse retraction of the 6 anterior teeth using temporary skeletal anchorage devices as the exclusive source of anchorage. No brackets or bands were placed on the posterior dentition during retraction. Regarding the lingual group, the mean change in the upper incisor inclination to SN plane of 7.8 degrees, with a standard deviation of 5.5 was reported by Kim et al who compared pre-treatment cephalometric radiographs with those taken after en-masse retraction of the 6 anterior teeth using the lingual biocreative therapy technique.

The effect size ratio was calculated to be 1.212 using G*power software (Universität Düsseldorf, Germany). A t-test assuming equal variance for two independent groups was used and the power was set as 0.8, allocation ratio of 1:1 and the Type I error probability (alpha) associated with this test was set as 0.05. Results of the test showed that "the group sample sizes of 12 each would achieve 80.09% power to reject the null hypothesis of equal means with a significance level (alpha) of 0.05 using a two-sided two-sample equal variance t-test".

Therefore, 24 subjects will be needed, with 12 subjects in each group. To account for patient loss to follow up (attrition), a sample size of 30 patients will be selected and divided into two groups, fifteen each.

7b. Interim analysis and stopping guidelines In both groups, in case of mobility in the skeletal anchorage device used in any subject, the load will be removed for about two weeks and oral hygiene instructions will be reinforced. After that, the load will be restored. If the mobility persists, surgical exposure of the skeletal anchorage device will be done and either insertion of longer mini screws or a change in the position of the skeletal anchorage device will be done.

Any harms, adverse effects or unintended effects of the study intervention will be documented and reported. Post-surgical swelling and pain are anticipated and will be addressed by antibiotics and pain killers. Other unanticipated surgical harms have to be immediately managed and will be reported. Harms related to the orthodontic appliances will be managed by the principal investigator.

8. Randomization 8a. Sequence generation The randomization of the recruited subjects will be done with a randomized list, using random.org website. This list is made by an individual not involved in the clinical trial (A.Z.) 8b. Type The type of randomization will be block randomization. The number of blocks and block size will be blinded to the investigators.

9. Allocation and concealment mechanism

* Each patient will be allocated a number from sequentially numbered opaque sealed envelopes after fulfilment of the inclusion criteria and signing the informed consent to be enrolled in the study.
* According to the number, the patients will be then allocated into one of the groups using a randomization table.

  10. Implementation Before the beginning of the research, the allocation sequence will be generated by a person not involved in the study (Dr A.Z.). The random list will be sealed from the principal investigator who will enrol participants. After the participant takes a sealed number, A.Z. will be contacted to implement the allocation. All the study contributors will have no access to the random list. The envelopes will be closed with the type of treatment selected for storage of the information.

  11. Blinding Blinding will be carried out only for the data assessment because the researchers, participants and subjects can not be blinded. Therefore, a person who does not know the nature of the trial will analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Full permanent dentition (excluding third molars)
* Angle class II malocclusion with increased overjet. Treatment plan includes extraction of the upper first premolars and retraction of the maxillary anterior teeth with maximum anchorage.

Exclusion Criteria:

* • Systemic diseases (examples include bleeding disorders, bisphosphonate therapy, chemotherapy, and radiotherapy) or craniofacial anomaly.

  * Previous orthodontic treatment.
  * Obvious periodontal disease and signs of bone loss.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-17 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Type of anterior tooth movement. | Expected average of 10 months
  This would be detected by measurement of the mean change in bucco-lingual inclination of every anterior tooth from the baseline. This outcome will be measured after achieving a normal overjet.

SECONDARY OUTCOMES:
Change in the nasolabial angle. | Expected average of 10 months
  Measurement of the mean change in nasolabial angle
Molar anchorage loss | Expected average of 10 months
  Measurement of the mean change in the antero-posterior position of the first molar crown
Patient satisfaction from treatment with either the labial or lingual biocreative therapy | Expected average of 10 months
  Detected by using a questionnaire filled by the patients at the end of the retraction period
Changes in the transverse dimension of the upper arch. | Expected average of 10 months
  Detected through measurement of the mean change of the inter-canine and inter-molar width from the baseline
Vertical movement of the crown of the six maxillary anterior teeth | Expected average of 10 months
  Detected by measurement of the mean change in the vertical linear distance from the incisal edge/cusp tip of every tooth to the palatal plane
point A to Nasion perp plane | Expected average of 10 months
  Measurement of the mean change in the position of point A from the Nasion perpendicular plane
Time duration required to complete the retraction phase. | Expected average of 10 months
  Recorded in months and days, from the start till the end of retraction period
change in inter-labial gap | Expected average of 10 months
  Measurement of the mean change in inter-labial gap
upper lip position | Expected average of 10 months
  Change in the position of the upper lip in the antero-posterior dimension
Lower lip position | Expected average of 10 months
  Change in the position of the lower lip in the antero-posterior dimension

CONTACTS AND LOCATIONS:
Overall Officials: Mais M Sadek, MSc, Principal Investigator — Associate lecturerof Orthodontics, Ain Shams University; Noha E Sabet, PhD, Study Chair — Professor and Head of Orthodontic Department, Ain Shams University; Islam T Hassan, PhD, Study Director — Professor of Orthodontics, Ain Shams University

REFERENCES:
- [Background] Upadhyay M, Yadav S, Nagaraj K, Patil S. Treatment effects of mini-implants for en-masse retraction of anterior teeth in bialveolar dental protrusion patients: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2008 Jul;134(1):18-29.e1. doi: 10.1016/j.ajodo.2007.03.025. PMID 18617099
- [Background] Chung KR, Cho JH, Kim SH, Kook YA, Cozzani M. Unusual extraction treatment in Class II division 1 using C-orthodontic mini-implants. Angle Orthod. 2007 Jan;77(1):155-66. doi: 10.2319/020106-35R.1. PMID 17029536
- [Background] Chung KR, Kim SH, Kook YA, Son JH. Anterior torque control using partial-osseointegrated mini-implants: biocreative therapy type I technique. World J Orthod. 2008 Summer;9(2):95-104. PMID 18575303
- [Background] Chung KR, Kim SH, Kook YA, Choo H. Anterior torque control using partial-osseointegrated mini-implants: biocreative therapy type II technique. World J Orthod. 2008 Summer;9(2):105-13. PMID 18575304
- [Background] Su J, Liu J, Zhang D, Luo G, Chen L, Yu X, Lin Z, Zhang J. [Finite-element investigation on center of resistance of maxillary anterior teeth]. Sheng Wu Yi Xue Gong Cheng Xue Za Zhi. 2014 Oct;31(5):994-1000. Chinese. PMID 25764710
- [Background] Miyawaki S, Yasuhara M, Koh Y. Discomfort caused by bonded lingual orthodontic appliances in adult patients as examined by retrospective questionnaire. Am J Orthod Dentofacial Orthop. 1999 Jan;115(1):83-8. doi: 10.1016/s0889-5406(99)70320-3. PMID 9878962
- [Background] Hong RK, Heo JM, Ha YK. Lever-arm and mini-implant system for anterior torque control during retraction in lingual orthodontic treatment. Angle Orthod. 2005 Jan;75(1):129-41. doi: 10.1043/0003-3219(2005)0752.0.CO;2. PMID 15747828
- [Background] Park YC, Choi YJ, Choi NC, Lee JS. Esthetic segmental retraction of maxillary anterior teeth with a palatal appliance and orthodontic mini-implants. Am J Orthod Dentofacial Orthop. 2007 Apr;131(4):537-44. doi: 10.1016/j.ajodo.2005.05.051. PMID 17418722
- [Background] Kim JS, Kim SH, Kook YA, Chung KR, Nelson G. Analysis of lingual en masse retraction combining a C-lingual retractor and a palatal plate. Angle Orthod. 2011 Jul;81(4):662-9. doi: 10.2319/100110-574.1. Epub 2011 Mar 14. PMID 21406002
- [Background] Kim SH, Hwang YS, Ferreira A, Chung KR. Analysis of temporary skeletal anchorage devices used for en-masse retraction: a preliminary study. Am J Orthod Dentofacial Orthop. 2009 Aug;136(2):268-76. doi: 10.1016/j.ajodo.2007.08.023. PMID 19651358
- [Derived] Sadek MM, Sabet NE, Hassan IT. Type of tooth movement during en masse retraction of the maxillary anterior teeth using labial versus lingual biocreative therapy in adults: A randomized clinical trial. Korean J Orthod. 2019 Nov;49(6):381-392. doi: 10.4041/kjod.2019.49.6.381. Epub 2019 Nov 26. PMID 31815106